CLINICAL TRIAL: NCT06752486
Title: Assessment of Safety and Efficacy of Gabapentin for Postoperative Analgesia After Surface Ablation, Versus Diclofenac Potassium as a Gold Standard
Brief Title: Assessment of Safety and Efficacy of Gabapentin After Surface Ablation, a Case Control Experimental Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Research Institute of Ophthalmology, Egypt (Other)
Responsible Party: Principal Investigator, Dina Moustafa Mohamed, Principal investigator, Research Institute of Ophthalmology, Egypt
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-2-23-3-6
Record Dates: First submitted 2024-12-15; First posted 2024-12-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Pain After Photorefractive Keratectomy; VAS Will be Used to Assess Pain Postoperative
MeSH Terms: interventions — Analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gabapentin Group (Active Comparator): The first group will be given gabapentin orally in a dose of 300mg three times daily post photorefractive keratectomy for 72 hours
  Interventions: Drug: Giving post photorefractive keratectomy for pain relief
- Diclofenac potassium Group (Active Comparator): the second group will be given oral diclofenac potassium 50mg Tid for 72 hours. The drugs will be administered starting from the first day postoperative.
  All patients will be subjected to:
  1. History taking including sociodemographics, medical illnesses, and prior surgery or anesthetic experiences.
  2. Examination including assessment of vital data (heart rate, blood pressure, respiratory rate, level of consciousness, and respiratory examination.
  Interventions: Drug: Giving post photorefractive keratectomy for pain relief

INTERVENTIONS:
Drug: Giving post photorefractive keratectomy for pain relief — We plan to conduct a randomized prospective study to assess the efficacy and safety of oral Gabapentin versus oral Diclofenac Potassium for postoperative analgesia in adults undergoing surface ablation. The first group will be given gabapentin orally in a dose of 300mg Tid for 72 hours and the second group will be given oral diclofenac potassium 50mg Tid for 72 hours. The drugs will be administered starting from the first day postoperative.

SUMMARY:
The current study aims at assessing the efficacy and safety of oral Gabapentin alone versus Diclofenac Potassium drugs for postoperative analgesia in patients undergoing surface ablation.

DETAILED DESCRIPTION:
To estimate the analgesic effect and pain severity after surface ablation with oral Gabapentin intake in comparison with Diclofenac Potassium, where Gabapentin could be a better analgesic medication after surface ablation

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years old
* preoperative stable refraction for at least one-year,
* normal corneal tomography with expected postoperative flat K reading not less than 38D, and postoperative residual stromal bed not less than 350 μm.

Exclusion Criteria:

* Patients with preoperative corrected distance visual acuity (CDVA) of worse than 20/30
* amblyopic patients,
* patients with a history of previous ocular surgeries,
* herpetic eye infection, or corneal dystrophies.
* Patients with other ocular conditions e.g. uveal or retinal diseases, and glaucoma
* Diabetics,
* Hypertensives,
* Kidney problems,
* breathing problems
* Adults older than 65 years.
* Previous allergy or adverse reaction to the used drugs.
* History of drug abuse or alcohol abuse problems
* History of mood problems, depression suicidal thoughts or behavior

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative Pain intensity will be evaluated with the visual analog scale (VAS) after surgery up to 72 hours. | 72 hours postoperative
  pain assessment using Visual Analogue Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of Ophthalmolgy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
patient privacy